CLINICAL TRIAL: NCT04152733
Title: Effect of High Flow Nasal Cannula on Oxygenation During Urodynamic Study in Pediatric Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H1910-038-1068
Record Dates: First submitted 2019-11-03; First posted 2019-11-05 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Desaturation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Children in the control group receive oxygen via conventional nasal cannula during deep sedation. Oxygen flow is determined to set the fraction of inspired oxygen of 50%.
- High flow (HF) group (Experimental): Children in the HF group receive oxygen via high flow nasal cannula during deep sedation. Fraction of inspired oxygen is set to 50%.
  Interventions: Device: High flow nasal cannula

INTERVENTIONS:
Device: High flow nasal cannula — Oxygen is supplied via high flow nasal cannula. Heated air (2L/kg/min) is administered using Optiflow device (Fisher and Paykel Healthcare, Auckland, New Zealand).
  Arms: High flow (HF) group

SUMMARY:
To evaluate the effect of high flow nasal cannula for prevention of hypoxia during deep sedation in pediatric population

ELIGIBILITY:
Inclusion Criteria:

* Children aged <7 years
* ASA class I, II

Exclusion Criteria:

* Respiratory disease
* Pneumothorax
* Increased ICP
* Nasal bleeding
* Previous airway surgery
* Trauma
* Pulmonary hypertension

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Estimated)
Dates: Start 2020-03-23 (Actual); Primary Completion 2021-11-20 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of desaturation | During deep sedation (during approximately 1 hour after propofol infusion)
  Incidence of peripheral pulse oximeter value lower than 95%

SECONDARY OUTCOMES:
Minimum pulse oximeter value | During deep sedation (during approximately 1 hour after propofol infusion)
Incidence of peripheral pulse oximeter value lower than 90% | During deep sedation (during approximately 1 hour after propofol infusion)
Incidence of changes in oxygen flow (control group) or FiO2 (HF group) | During deep sedation (during approximately 1 hour after propofol infusion)
percutaneous CO2 value | During deep sedation (during approximately 1 hour after propofol infusion)
Oxygen reserve index value | During deep sedation (during approximately 1 hour after propofol infusion)
Incidence of manual ventilation | During deep sedation (during approximately 1 hour after propofol infusion)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No